CLINICAL TRIAL: NCT01320683
Title: A Phase II Trial of Radioimmunotherapy (Y-90 M5A) Following Hepatic Resection and FOLFIRI or FOLFOX Chemotherapy [+/-BEVACIZUMAB], or Xelox for Metastatic Colorectal Carcinoma to the Liver
Brief Title: Combination Chemotherapy and Bevacizumab Before Surgery and Radiolabeled Monoclonal Antibody Therapy in Treating Liver Metastases in Patients With Metastatic Colorectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual.
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09053; NCI-2011-00369 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P01CA043904 (NIH)
Record Dates: First submitted 2011-03-18; First posted 2011-03-22 (Estimated); Results first posted 2016-06-20 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-06

CONDITIONS: Liver Metastases; Recurrent Colon Cancer; Recurrent Rectal Cancer; Stage IVA Colon Cancer; Stage IVA Rectal Cancer; Stage IVB Colon Cancer; Stage IVB Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Oxaliplatin; Leucovorin; Fluorouracil; Bevacizumab; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (combination chemotherapy and radioimmunotherapy) (Experimental): FOLFOX* + BEVACIZUMAB CHEMOTHERAPY: Patients receive oxaliplatin IV over 2 hours, leucovorin calcium IV over 2 hours, fluorouracil IV continuously over 46-48 hours, and bevacizumab IV over 30-90 minutes. Treatment repeats for up to 12 courses in the absence of disease progression or unacceptable toxicity. RIT: Within 4-12 weeks after completion of post-hepatic resection therapy chemotherapy, patients receive yttrium Y 90 DOTA anti-CEA monoclonal antibody M5A IV over 25 minutes. Treatment repeats every 6-10 weeks for 2 courses in the absence of disease progression or unacceptable toxicity. NOTE:*Patients previously failing oxaliplatin regimen receive FOLIFIRI chemotherapy comprising irinotecan hydrochloride IV over 90 minutes, leucovorin calcium over 2 hours, fluorouracil IV continuously over 46-48 hours, and bevacizumab IV over 30-90 minutes. Treatment repeats for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: oxaliplatin; Drug: leucovorin calcium; Drug: fluorouracil; Biological: bevacizumab; Radiation: yttrium Y 90 DOTA anti-CEA monoclonal antibody M5A; Other: laboratory biomarker analysis; Other: pharmacological study; Drug: irinotecan hydrochloride

INTERVENTIONS:
Drug: oxaliplatin — Given IV
  Other Names: 1-OHP; Dacotin; Dacplat; Eloxatin; L-OHP
Drug: leucovorin calcium — Given IV
  Other Names: CF; CFR; LV
Drug: fluorouracil — Given IV
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF
Radiation: yttrium Y 90 DOTA anti-CEA monoclonal antibody M5A — Given IV
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Drug: irinotecan hydrochloride — Given IV
  Other Names: Campto; Camptosar; CPT-11; irinotecan; U-101440E

SUMMARY:
This phase II trial studies how well giving combination chemotherapy and bevacizumab before surgery and radiolabeled monoclonal antibody therapy works in treating liver metastases in patients with metastatic colorectal cancer. Drugs used in chemotherapy, such as leucovorin calcium, fluorouracil, and oxaliplatin (FOLFOX), work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Radiolabeled monoclonal antibodies, such as yttrium Y 90 DOTA anti-CEA monoclonal antibody M5A, can find tumor cells and carry tumor-killing substances to them without harming normal cells. Giving chemotherapy and monoclonal antibody before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving radiolabeled monoclonal antibody therapy after surgery may kill any tumor cells that remain after surgery

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the progression free survival in colorectal cancer patients after hepatic resection of liver metastases and FOLFOX or leucovorin calcium, fluorouracil, and irinotecan hydrochloride (FOLFIRI) chemotherapy [+/- Bevacizumab], or capecitabine and oxaliplatin (XELOX),followed by intravenous (IV) yttrium-90 (90Y) M5A anti-CEA antibody.

SECONDARY OBJECTIVES:

I. To study the feasibility and toxicities of such adjuvant therapy following resection and/or ablation of liver metastases and FOLFOX chemotherapy.

II. To evaluate the biodistribution, clearance and metabolism of 90Y and 111In (indium-111) M5A administered IV.

OUTLINE:

FOLFOX* + BEVACIZUMAB CHEMOTHERAPY: Patients receive oxaliplatin IV over 2 hours, leucovorin calcium IV over 2 hours, fluorouracil IV continuously over 46-48 hours, and bevacizumab IV over 30-90 minutes. Treatment repeats for up to 12 courses in the absence of disease progression or unacceptable toxicity.

RADIOIMMUNOTHERAPY (RIT): Within 4-12 weeks after completion of post-hepatic resection therapy chemotherapy, patients receive yttrium Y 90 DOTA anti-CEA monoclonal antibody M5A IV over 25 minutes. Treatment repeats every 6-10 weeks for 2 courses in the absence of disease progression or unacceptable toxicity.

NOTE:*Patients previously failing oxaliplatin regimen receive FOLIFIRI chemotherapy comprising irinotecan hydrochloride IV over 90 minutes, leucovorin calcium over 2 hours, fluorouracil IV continuously over 46-48 hours, and bevacizumab IV over 30-90 minutes. Treatment repeats for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a Karnofsky performance status of >= 60%
* Patients must have histological confirmation of colorectal carcinoma
* Patients must have colorectal tumors that produce carcinoembryonic antigen (CEA) as documented by either immunohistochemistry or by an elevated serum CEA
* Patients will be enrolled on this trial after resection of hepatic metastases combined with FOLFIRI or FOLFOX [+/- Bevacizumab], or XELOX; patients may have received a maximum of 12 cycles of FOLFIRI or FOLFOX [+/- Bevacizumab], or XELOX, which includes chemotherapy prior to and post hepatic resection
* Prior radiotherapy, immunotherapy, or chemotherapy must have been completed between 4-12 weeks prior to patient entry on this study and patients must have recovered from all expected acute side effects of the prior therapy
* Hemoglobin >= 10 gm %; patients may be transfused to reach a hemoglobin >= 10 gm %
* White blood cell (WBC) >= 4000/uL
* Absolute neutrophil count (ANC) >= 1,500/mm^3
* Platelets >= 150,000/ul
* Patients may have history of prior malignancy for which the patient has been disease-free for five years; basal or squamous cell skin cancers or carcinoma in situ of the cervix are allowed regardless of diagnosis date
* Patients must have no prior history of radiation therapy to the liver (includes 90Y microsphere therapy)
* Patients must have a total bilirubin =< 1.5 mg/dL
* Serum creatinine of =< 1.5 x upper limit of normal (ULN)
* Patients must have had < 40% liver resected at the close of completion of the hepatic resection; this will be verified retrospectively
* Serum human immunodeficiency virus (HIV) testing and hepatitis B surface antigen and hepatitis C antibody testing must be negative
* Women of childbearing potential must have a negative serum pregnancy test prior to entry and while on study must be practicing an effective form of contraception
* If a patient has previously received murine or chimeric antibody, then serum anti-antibody testing must be negative
* Computed tomography (CT) scan restaging done prior to RIT must demonstrate no evidence of progressive disease
* The patient must be seen in consultation by the radiation oncologist who will be administering the radiolabeled antibody therapy and must be informed of the potential risks and side effects of the therapy, and informed consent must be documented in the consultation note

Exclusion Criteria:

* Patients that have received radiation therapy to greater than 50% of their bone marrow
* Patients with any nonmalignant intercurrent illness (example cardiovascular, pulmonary, or central nervous system disease) which is either poorly controlled with currently available treatment or which is of such severity that the investigators deem it unwise to enter the patient on protocol shall be ineligible
* Chronic active hepatitis, cirrhosis, or chemotherapy steatohepatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Wong, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Combination Chemotherapy and Radioimmunotherapy)
Started | 1
Completed | 0
Not Completed | 1
Not completed — Positive antibody response | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Combination Chemotherapy and Radioimmunotherapy)
Number analyzed (Participants) | 1
Age, Continuous [Median (Full Range); unit: years] | 66 [66 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Estimated using the product-limit method of Kaplan-Meier, and 95% confidence limits calculated for these estimates.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Up to 24 months
Arm/Group | Treatment (Combination Chemotherapy and Radioimmunotherapy)
Number analyzed (Participants) | 0

2. Secondary Outcome: Overall Survival
Description: Overall Survival is calculated for all patients from the date of initial treatment to date of death due to any cause. Patients who were still alive were censored at the date of last follow-up. Survival rates were estimates using the Kaplan-Meier method, and 95% confidence limits calculated for these estimates.
Time Frame: Up to 5 years
Arm/Group | Treatment (Combination Chemotherapy and Radioimmunotherapy)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events occurred over a two month period
Description: All adverse events are included regardless of grade and attribution.
Arm/Group | Treatment (Combination Chemotherapy and Radioimmunotherapy)
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Combination Chemotherapy and Radioimmunotherapy) (N=1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
INR increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vaginal dryness (Reproductive system and breast disorders) | 1 (1)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1)
Weight gain (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination due to slow accrual. Unable to perform planned analysis due to the small number of subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes